CLINICAL TRIAL: NCT00142116
Title: Phase II Study of Thalidomide and Rituximab in Waldenstrom's Macroglobulinemia
Brief Title: Thalidomide and Rituximab in Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven P. Treon, MD, PhD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Cape Cod Hospital (Other)
Responsible Party: Sponsor-Investigator, Steven P. Treon, MD, PhD, Director, Bing Center for WM, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-077
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Waldenstrom's Macroglobulinemia; Lymphoplasmacytic Lymphoma
Keywords: thalidomide; rituximab; Waldenstrom's
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Thalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide and Rituximab (Experimental): Thalidomide 200mg orally once a day for 14 weeks if that dosage is tolerated well, it will be increased to 400mg for up to 50 weeks
  Rituximab Given intravenously once weekly for 4 weeks beginning the second week of study treatment. If tolerated well, this may be repeated 8 weeks later.
  Interventions: Drug: Thalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Thalidomide — 200mg orally once a day for 14 weeks if that dosage is tolerated well, it will be increased to 400mg for up to 50 weeks.
  Other Names: Thalomid
Drug: Rituximab — Given intravenously once weekly for 4 weeks beginning the second week of study treatment. If tolerated well, this may be repeated 8 weeks later.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the percentage of people who can attain remission and the length of time such responses to therapy are sustained, as well as the side effects that might result from rituximab and thalidomide in people with lymphoplasmacytic lymphoma.

DETAILED DESCRIPTION:
* Patients will receive thalidomide(200mg) orally once daily for two weeks. If after two weeks of thalidomide, the patient is doing well the dose of thalidomide will increase (400mg) and they will remain on it for up to 50 additional weeks. The length of time a patient is on thalidomide will depend upon how they are responding to therapy.
* During the second week of the study patients will also begin receiving rituximab intravenously once weekly for 4 weeks, which may then be repeated 8 weeks later depending upon the response.
* A determination of how the patient is responding will be made based on testing conducted at 12 weeks. This testing includes blood tests and possibly a bone marrow biopsy. If it is determined that the disease is not progressing, patients will begin a second phase of treatment which includes 4 additional weekly infusions of rituximab and the continuation of oral thalidomide.
* If it is determined at the 12-week evaluation, or at any time thereafter, that the disease has progressed (by studying serum immunoglobulin M (IgM) levels, bone marrow involvement, tumor cells, and/or development of new signs and symptoms) then the patient will be removed from the study.
* Periodic examinations and tests will be done to determine how the patient is doing, what response and side effects (if any) the patient may be having from the study drugs. If patient is responding to therapy then they will remain on this study and followed for a period of two years.
* Bone marrow biopsies and aspirations will be obtained at 3-6 month intervals extending for 2 years following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia requiring therapy
* Baseline staging requirements
* Absolute Neutrophil Count > 500/microliter (uL)
* Platelet Count > 25,000/uL
* Serum creatinine < 2.5mg/dL
* Total bilirubin and transaminase (SGOT) < 2.5 X Upper Limit of Normal (ULN)
* Greater than 18 years of age
* Life expectancy of 3 months or greater
* Eastern Cooperative Oncology Group (ECOG) status performance of 0-2

Exclusion Criteria:

* Chemotherapy, steroid therapy, or radiation therapy within 30 days of study entry
* Pregnant or lactating women
* Serious co-morbid disease
* Uncontrolled bacterial, fungal or viral infection
* Active second malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-05; Primary Completion 2004-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Result] Treon SP, Soumerai JD, Branagan AR, Hunter ZR, Patterson CJ, Ioakimidis L, Briccetti FM, Pasmantier M, Zimbler H, Cooper RB, Moore M, Hill J 2nd, Rauch A, Garbo L, Chu L, Chua C, Nantel SH, Lovett DR, Boedeker H, Sonneborn H, Howard J, Musto P, Ciccarelli BT, Hatjiharissi E, Anderson KC. Thalidomide and rituximab in Waldenstrom macroglobulinemia. Blood. 2008 Dec 1;112(12):4452-7. doi: 10.1182/blood-2008-04-150854. Epub 2008 Aug 19. PMID 18713945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Waldenstrom's Macroglobulinemia
Pre-assignment Details: A phase II study using thalidomide and rituximab in symptomatic Waldenstrom's macroglobulinemia (WM) patients naïve to either agent.
Groups:
- All WM Patients: Waldenstrom's Macroglobulinemia Patients
Period: Overall Study
Arm/Group | All WM Patients
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All WM Patients
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Response determinations were made using modified consensus panel criteria from the Third International Workshop on WM, and response rates were determined on an evaluable basis. A complete response was defined as having resolution of all symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly. Patients achieving a partial response and a minor response were defined as achieving a more than or equal to 50% and more than or equal to 25% reduction in serum IgM levels, respectively. Patients with stable disease were defined as having less than 25% change in serum IgM levels, in the absence of new or increasing adenopathy or splenomegaly and/or other progressive signs or symptoms of WM. Progressive disease was defined as a greater than 25% increase in serum IgM level occurred from the lowest attained response value or progression of clinically significant disease-related symptom(s).
Time Frame: 3 years
Population: Intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | All WM Patients
Number analyzed (Participants) | 25
participants
  Complete Response | 1
  Partial Response | 15
  Minor Response | 2
  Stable Disease | 7

2. Secondary Outcome: To Identify the Mechanism(s) of Action for Combined Thalidomide and Rituximab Activity.
Time Frame: 3 years
Reporting Status: Not Posted

3. Primary Outcome: Time to Progression
Description: Time to disease progression (TTP) was calculated from the start of therapy using the Kaplan-Meier method.
Time Frame: 49.1 months
Measure: Median (Full Range); unit: months
Groups:
- Thalidomide and Rituximab: Thalidomide 200mg orally once a day for 14 weeks if that dosage is tolerated well, it will be increased to 400mg for up to 50 weeks
  Rituximab Given intravenously once weekly for 4 weeks beginning the second week of study treatment. If tolerated well, this may be repeated 8 weeks later.
  Thalidomide: 200mg orally once a day for 14 weeks if that dosage is tolerated well, it will be increased to 400mg for up to 50 weeks.
  Rituximab: Given intravenously once weekly for 4 weeks beginning the second week of study treatment. If tolerated well, this may be repeated 8 weeks later.
Arm/Group | Thalidomide and Rituximab
Number analyzed (Participants) | 25
months
  TTP for all evaluable patients | 34.8 [1.0 to 49.1]
  TTP for responding patients | 38.7 [10.3 to 49.1]
  TTP for previously treated patients | 15.25 [1.0 to 45.8]
  TTP for previously untreated patients | 36.04 [2.5 to 49.1]

ADVERSE EVENTS:
Arm/Group | All WM Patients
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All WM Patients (N=25)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — COPD Exacerbation with respiratory failure related to long standing smoking, not related to protocol therapy.
Death (Cardiac disorders) | 1 (1) — Sudden death in a patient with longstanding hypertensive disease and arthrosclerosis while playing golf.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All WM Patients (N=25)
Peripheral Neuropathy (Nervous system disorders) | 11 (11)
Somnolence (Nervous system disorders) | 3 (3)
Confusion (Nervous system disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Tremors (Nervous system disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No